CLINICAL TRIAL: NCT05502692
Title: A Cross-sectional, Observational Study to Characterise the Transition to Dolutegravir-based Regimens in South Africa in Terms of the Emergence of Obesity, Viral Re-suppression and Integration Into Routine Programme Care
Brief Title: CHARACTERISE - A Cross-sectional, Observational Study to Characterise the Transition to Dolutegravir-based Regimens in South Africa in Terms of the Emergence of Obesity, Viral Re-suppression and Integration Into Routine Programme Care
Acronym: CHARACTERISE
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: UNITAID (Other)
Responsible Party: Principal Investigator, Professor Francois Venter, Professor, University of Witwatersrand, South Africa
Other Study IDs: EZ-FV-030
Record Dates: First submitted 2022-07-19; First posted 2022-08-16 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Dolutegravir
Keywords: The ADVANCE clinical trial; weight gain; viral re-suppression; regimens
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — Serum chemistry: serum sodium, potassium, chloride, bicarbonate Liver function: total protein, albumin, total bilirubin, direct bilirubin, alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), lactate dehydrogenase (LDH) Renal function: urea, creatinine, estimated creatinine clearance (Cockcroft-Gault method) Lipid panel: total cholesterol, triglycerides, HDL, and LDL cholesterol glucose metabolism: plasma glucose, HbA1C HIV virological suppression: plasma HIV-1 RNA An additional plasma (50 mL) sample will be stored for possible future analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: ADVANCE patient cohort, who have been on the TLD state programme for more than one year
  Interventions: Behavioral: CHARACTERISE
- Cohort 2: Existing cohorts of patients initiating TLE (and subsequently switched to TEE) more than 9 years ago and who have since transitioned to TLD within the state programme for more than one year.
  Interventions: Behavioral: CHARACTERISE

INTERVENTIONS:
Behavioral: CHARACTERISE — Cohort 1 Cohort 2

SUMMARY:
The ADVANCE clinical trial compared three recommended first-line regimens two containing dolutegravir head-to-head and demonstrated virological non-inferiority at 48- and 96-weeks respectively1,2, paving the way for the mass- introduction of dolutegravir-containing regimens across low- and- middle-income countries.

The dolutegravir-containing regimens in ADVANCE were very well tolerated and demonstrated remarkable viral re-suppression in patients with viraemia when adherence measures were instituted, even in the presence of genotypically-documented resistance1,2. Across Africa, including South Africa, and in many other low- and middle-income countries, the combination of tenofovir disoproxil fumarate/lamivudine (or emtricitabine) /dolutegravir has been rolled out to millions of patients, much of this with Unitaid support to research, programmes and communities. Most ADVANCE patients have since transitioned out of the study and are on tenofovir disoproxil fumarate/lamivudine/dolutegravir in South African public sector clinics in central Johannesburg.

One of the unanticipated findings of ADVANCE and the concomitant Unitaid-supported NAMSAL3 study in Cameroon, as well as analyses of registration studies and observational studies, was the consistent finding that patients on dolutegravir experience significant weight gain and new-onset obesity. It remains unclear whether this is a feature of the integrase inhibitor class (and aggravated by tenofovir alafenamide), or whether other factors are at play - it is possible that HIV infection itself may predispose to weight gain in successfully treated patients, and other antiretrovirals may alter weight trajectories. The signal has been met with alarm by the public health community, as many countries where TLD is being rolled out are experiencing a parallel obesity epidemic. Obesity is strongly associated with adverse outcomes, including diabetes, cardio-vascular-disease (CVD), sleep apnoea, gastrointestinal and muscular-skeletal disorders, asthma, poor pregnancy outcomes, many cancers, mental health issues, and poor COVID-19 outcomes. In many countries with large antiretroviral programmes, these concurrent epidemics have significant public health and financial implications, and clarification of the extent of the obesity signal is urgent.

DETAILED DESCRIPTION:
This is a single centre, follow-up, observational, cross-sectional study reviewing two cohorts of patients who have transitioned to routine care on tenofovir disoproxil fumarate/lamivudine/dolutegravir . The first cohort will include ADVANCE patients, in which participants were randomised to one of three arms including either DTG+TAF/FTC, DTG+TDF/FTC or EFV/TDF/FTC. The second cohort will include patients previously on tenofovir disoproxil fumarate/lamivudine/emtricitabine or tenofovir disoproxil fumarate/emtricitabine/efavirenz who have since transitioned to routine care on tenofovir disoproxil fumarate/lamivudine/dolutegravir.

The medium 5-year data in the ADVANCE cohort and longer 9-year data in the other cohort metabolic and virologic consequences of those on long-term antiretrovirals will be described and compared in the above cohorts.

After obtaining informed consent from potential participants, a single cross-sectional, baseline visit will be conducted for each participant. Demographic data, clinical history, and details of previous and concomitant medications will be collected. Questionnaires including a food diary, Weight Bias Internalization Scale and Berlin questionnaire will be administered. Bone density and weight distribution will be assessed through use of a dual-energy X-ray absorptiometry DXA scan, and cardiac function assessed by conduction of a baseline electrocardiogram.

Laboratory evaluations will include a liver function test, glycated haemoglobin , plasma HIV-1 RNA viral load, lipid panel, C-peptide, both serum glucose and oral glucose tolerance test, and DNA extraction for genotyping in those with unsuppressed viral loads above 1000 copies/mL. Plasma samples will be stored locally for possible future analysis.

After the baseline visit, participants who are suitable for one, or more, sub-study will be identified. A randomly selected sub-group for each of the following sub-studies and additional investigations will be drawn from eligible participants within each cohort:

* Sleep evaluation: actigraphy and polysomnography
* Glucose metabolism evaluation: oral glucose tolerance test including assessment of glucose, insulin, and C-peptide to estimate insulin sensitivity and beta cell function
* Experiences of users and providers in the roll out of tenofovir disoproxil fumarate/lamivudine/dolutegravir in South Africa.

Abnormalities detected in the assessments will be managed by on-study medical personnel with referral as appropriate.

ELIGIBILITY:
Inclusion Criteria:

Adults of at least 18 years of age with HIV-1 infection who are currently on the TLD state programme who satisfy the below eligibility criteria.

The following eligibility criteria will be used to select study participants for the main study (baseline visit only):

* Inclusion criteria (baseline visit/main study):

  1. Able and willing to provide written or electronic informed consent for the baseline visit prior to any study-specific assessment or procedure.
  2. Age at least 18 years at the time of signing the informed consent form.
  3. Previously enrolled in the ADVANCE trial and have been on the TLD state programme for more than one year [Cohort 1] or, part of an existing cohort of patients initiating TLE (and switched to TEE) more than 9 years ago, who have been transitioned to TLD within the state programme for more than one year [Cohort 2].
  4. Access to a reliable telephone or other device permitting information transfer.

     Exclusion Criteria:
     * Exclusion criteria (baseline visit/main study):

  <!-- -->

  1. Personnel (e.g., investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study.
  2. Any physical, mental, or social condition, that, in the Investigator's judgment, might interfere with the completion of the baseline assessments and evaluations. The Investigator should make this determination in consideration of the volunteer's medical history.
  3. Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.

     Additional eligibility criteria will be used to identify study participants who are eligible for random selection for any of the sub-studies:
* Inclusion criteria (sub-studies):

  1. Enrolled into main study and completed baseline visit.
  2. Able and willing to provide written or electronic informed consent for the relevant sub-study.
  3. Identified as high risk for development of OSA based on the Berlin Questionnaire responses [Sleep sub study only].

Exclusion criteria (sub-studies):

1. Self-reported diabetic or on treatment for diabetes mellitus (Type 1 or 2) [Glucose metabolism sub-study only].
2. Serum glucose and/or HbA1C assessment at baseline consistent with a diagnosis of diabetes mellitus [Glucose metabolism sub-study only].

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two cohorts of patients who have transitioned to routine care on tenofovir disoproxil fumarate/lamivudine/dolutegravir (TLD). The first cohort will include ADVANCE patients, in which participants were randomised to one of three arms including either DTG+TAF/FTC, DTG+TDF/FTC or EFV/TDF/FTC. The second cohort will include patients previously on TLE or TEE who have since transitioned to routine care on TLD.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Characterisation of weight gain and metabolic consequences associated with long-term TLD use | 60 Days
  Weight measurement with body mass index calculation
Characterisation of weight gain and metabolic consequences associated with long-term TLD use | 60 Days
  Blood pressure which will measured using both systolic and diastolic
Characterisation of weight gain and metabolic consequences associated with long-term | 60 Days
  Plasma glucose
Characterisation of weight gain and metabolic consequences associated with long-term | 60 Days
  Oral glucose tolerance test
Characterisation of weight gain and metabolic consequences associated with long-term | 60 Days
  C-peptide measurements
Characterisation of weight gain and metabolic consequences associated with long-term | 60 Days
  Lipid panel
Characterisation of weight gain and metabolic consequences associated with long-term | 60 Days
  The liver function test will be performed to determine where damage may be occurring in the liver
Characterisation of weight gain and metabolic consequences associated with long-term | 60 Days
  Dual-energy X-ray absorptiometry (DXA) scan

SECONDARY OUTCOMES:
Assessment of factors contributing to, and individual perception on weight gain | 60 Days
  Food diary questionnaire there is no min and max values assessments will be done based upon participant diet
Assessment of factors contributing to, and individual perception on weight gain | 60 Days
  Weight Bias Internalization Scale through averaging 10 items (rated on a 1-7 scale), with higher scores indicating greater weight bias internalization
Description of the presence of viraemia | 60 Days
  Plasma HIV-1 RNA levels
Description of the presence and patterns of HIV-1 resistance mutations in participants with viral loads > 1000 copies/mL | 60 Days
  HIV-1 genotyping
Description and occurrence of associated sleep quality and disorders | 60 Days
  Berlin Questionnaire for risk of sleep apnoea
Description and occurrence of associated sleep quality and disorders | 60 Days
  Polysomnography in randomly selected 20% of participants at high risk of developing obstructive sleep apnoea based on the Berlin Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn Bosch, MBBCh, Principal Investigator — Ezintsha, a division of Wits Health Consortium
Locations (1):
- Sunnyside Office Park, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT05502692/Prot_SAP_000.pdf